CLINICAL TRIAL: NCT00183144
Title: A Therapeutic Workplace for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAASIL12154; R01AA012154 (NIH); NIH RO1 - AA12154
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2007-10

CONDITIONS: Alcohol Dependence
Keywords: contingency management; reinforcement; employment; Therapeutic Workplace
MeSH Terms: conditions — Alcoholism

INTERVENTIONS:
Behavioral: Contingency management

SUMMARY:
The purpose of this study is to determine whether the Therapeutic Workplace is effective in increasing and maintaining long-term drug abstinence in homeless, alcohol dependent adults.

DETAILED DESCRIPTION:
Few populations are beset with the constellation of economic, social and health problems that afflict homeless individuals. At the heart of much of this misfortune are staggering rates of alcoholism and drug addiction. While it is not clear whether substance abuse is a cause, consequence, or simply a correlate of homelessness, there is no question that substance abuse is among the most common and most serious problems facing the homeless. Given their unique set of serious and chronic problems, the Institute of Medicine has identified the homeless as a group of people in need of specialized substance abuse interventions. Prior research has shown that the Therapeutic Workplace intervention is effective in the treatment of chronically unemployed heroin and cocaine dependent individuals. The intervention integrates abstinence reinforcement contingencies of proven efficacy into a model supported work program. Under this intervention, patients are paid to perform data entry jobs in the Therapeutic Workplace. Those lacking needed skills are given intensive training in basic academic and job skills. To reinforce abstinence from alcohol and drugs, patients are required to provide an alcohol-free breath sample and drug-free urine sample to gain entrance to the workplace each day. In this way, patients can work and earn salary only when they abstain from alcohol and drugs. Patients are paid in vouchers instead of cash to reduce the chance they will use their earnings to purchase alcohol or drugs.

A randomized trial was conducted to evaluate the efficacy of this intervention in homeless, alcohol-dependent adults who completed an inpatient alcohol detoxification. After the detoxification, 124 participants were invited to attend the workplace for 6 months. They were randomly assigned to one of three groups that differed in the requirements for voucher reinforcement. One group received the full therapeutic workplace intervention in which vouchers were contingent on both abstinence and work (Abstinence and Work group). A second group was paid for work, but did not have to provide an alcohol-free breath sample or drug-free urine sample to gain access to the workplace; their vouchers were contingent on work only (Work-Only group). A third group was invited to attend the therapeutic workplace but received no vouchers for work performed or abstinence achieved during treatment (No Voucher group).

ELIGIBILITY:
Inclusion Criteria:

* meet DSM IV criteria for alcohol dependence
* are homeless in that they lack a fixed nighttime residence
* are unemployed
* are at least 18 years old

Exclusion Criteria:

* are currently physically dependent on opioids
* are considered in imminent risk of suicide
* have a psychiatric disorder that is likely to result in behaviors that could disrupt the workplace functioning or limit their ability to provide informed consent
* are physically unable to perform typing or keypad entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156
Dates: Start 2001-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
percentage of 30 day assessments that subjects reported alcohol abstinence
percentage of heavy drinking days
percentage of positive breath-alcohol tests
percent of patients meeting criteria for current alcohol dependence

SECONDARY OUTCOMES:
percentage of urine samples negative for other drugs
percentage of participants employed each month
days employed per month
employment income per month

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, PhD, Principal Investigator — Johns Hopkins/Center for Learning and Health
Locations (1):
- Center for Learning and Health, Johns Hopkins Bayview Medical Campus, 5200 Eastern Ave., Suite W142, Baltimore, Maryland, United States